CLINICAL TRIAL: NCT07156994
Title: Unravelling Health and Frequent Symptoms and Voice Characteristics Evolution Over Time of Users of the Long COVID Companion Application to Develop Voice Biomarkers of Frequent Long Covid-related Symptoms
Brief Title: Development of Voice Biomarkers of Frequent COVID-19 and Long Covid-related Symptoms Based on Data From Users of the Long COVID Companion App
Acronym: EVO-LC
Status: Not yet recruiting | Type: Observational
Sponsor: Luxembourg Institute of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: EVO-LC
Record Dates: First submitted 2025-09-02; First posted 2025-09-05 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-08

CONDITIONS: Long COVID
Keywords: Long COVID; Vocal biomarkers; symptoms
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long Covid Companion (LCC) app users: Study participation will consist in a follow-up of maximum 36 months after the signature of the electronic informed consent form. The participants will be invited to use the app in the manner they want, in terms of frequency and functionalities used.
  Participants who were already using the app before signing the study informed consent form will be asked if they agree to the use of the data previously collected between the account creation and the informed consent signature for the study.
  In addition, study participants will be invited to do regular standardized voice recordings (at the same time as their regular health evaluation) and to complete the symptom questionnaires at the same time. Very short questions (Ecological Momentary Assessments), followed by one standardized voice recording, will also be sent during the first 8 days after signature of the study informed.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — Participants will be followed digitally using the LCC app. They will complete questionnaires about their health status and do voice recordings on their own rhythm during the entire study duration.

SUMMARY:
The LIH DDP research team focuses its research topics on vocal biomarkers and Long COVID, among others. Voice is indeed a promising tool to monitor health, as it contains many information on our health and is easy to collect.

The development of vocal biomarkers of Long COVID-related symptoms could improve the remote monitoring of the health status of people affected by this disease.

The LIH developed the Long COVID Companion (LCC) app in collaboration with the ApresJ20 Long COVID patient association in France to support patients in their daily lives. LCC app users will be invited to participate in this study to collect voice recordings at the same time as health-related data.

The objectives of this study are:

Primary objective: To develop vocal biomarker candidates for the main Long COVID symptoms (fatigue, brain fog, respiratory problems, sleep issues, stress, anxiety,..) in a population of people with Long COVID.

Secondary objectives:

* to assess the intra-individual longitudinal evolution of voice characteristics of people with LC
* to assess app usability and acceptability in the long-term.

DETAILED DESCRIPTION:
Five years after the start of the COVID-19 pandemic, it has been estimated that a mean of 10-20% of COVID-19 patients will develop Long COVID, which represents at least 65 million people worldwide. In Luxembourg, based on the current status of the COVID-19 pandemic and the prevalence of Long COVID in other countries, we estimate that approximately 25,000 individuals may have been affected by Long COVID.

People with Long COVID (PWLC) present complaints such as tachycardia, extreme fatigue, dyspnea, and inability to perform daily physical tasks. More than 200 symptoms have been associated with Long COVID, and multiple organs are affected. Our previous work showed that 59% of COVID-19-infected people from the PrediCOVID cohort study reported 1 or more persisting symptom(s) after one year. The number of persisting symptoms increased with the initial disease severity, and the quality of life of those participants was notably impacted by sleep disorders (54%) and compromised respiratory function (12.9%). Nonetheless, individuals with an initially asymptomatic or mild form of COVID-19 infection could also be affected.

Long COVID care, as for other chronic diseases, should align with the concept of minimally disruptive medicine, aiming for a reduced burden on patients' lives while maximizing health outcomes. PWLC frequently have several healthcare professionals in charge of different aspects of their care, with many appointments and travels to manage. They are also regularly asked to complete long standardized questionnaires or scales to evaluate their symptoms, which generates an avoidable burden on their lives if care is not coordinated. The development of innovative methods to integrate multiple Patient Report Outcomes in a portable, versatile way, to reduce travels for medical care, and overall for remote health's monitoring is therefore of the highest importance.

Few existing apps that could meet the needs of PWLC already exist, such as "Visible" or "Living With". However, these apps are only available in the US and in the UK, respectively. Furthermore, the "Living with" app is available only by invitation. This limits their availability for PWLC in Europe. Some other apps designed for other chronic conditions, like myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS) Pacing app, are also used by some PWLC to manage their daily energy levels. However, these apps do not fully meet the specific needs of PWLC, and are only available in specific countries, in English, and some of them only on the iOS operating system, which restricts their potential use.

Voice is a promising candidate increasingly used in mobile health (mHealth) interactions in chronic diseases. Voice is an easy and cheap medium to collect and can be easily integrated into a device like a smartphone, now widely used by people of different ages and education levels. It can be used for vocal biomarker assessment as new clinical endpoints for relevant symptoms. Vocal biomarker candidates have already been identified by the Deep Digital Phenotyping (DDP) research team, based on data from the PrediCOVID cohort study, with performances above 80% to detect fatigue, loss of taste and smell, and symptomatic status in COVID-19-infected people. However, further progress is required before these vocal biomarkers can be used in clinical practice. New vocal biomarkers of global health status or of other symptoms need to be developed to allow a more personalized monitoring of PWLC.

The LIH developed the Long COVID Companion app based on the results of UpcomingVoice co-design study and in collaboration with the ApresJ20 Long COVID patient association in France. The app is the result of a participative process involving patients and healthcare professionals in charge of PWLC patients. App users can monitor their health and symptoms on a daily basis or at the frequency they want. App also offers the possibility to complete a daily life and a medical diary, a voice journaling, and to generate PDF reports with graphical visualization of symptom evolution. A new module dedicated to research with standardized voice recordings has been integrated in the app for the users who will take part in the present study The app was released in April 2024 and has more than 1700 users as of the end of March 2025.

It is of highest importance to assess the evolution of health of PWLC for a better understanding of the disease. Results will allow the development of personalized monitoring strategies by identifying vocal biomarkers of Long COVID symptoms and of the global health of PWLC.

As fatigue is the most frequent and impairing symptom of PWLC it is crucial to better understand the drivers of fatigue and to develop monitoring strategies.

The objectives of this study are :

Primary objective: To develop vocal biomarker candidates for the main Long COVID symptoms (fatigue, brain fog, respiratory problems, sleep issues, stress, anxiety,..) in a population of people with Long COVID.

Secondary objectives:

* to assess the intra-individual longitudinal evolution of voice characteristics of people with LC
* to assess app usability and acceptability in the long-term.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old)
* Male or female
* People with persisting symptoms related to COVID-19 (With Long COVID diagnosis or not)
* Adequate understanding of one of the study languages (English, French, German)
* Electronically signed informed consent form

Exclusion Criteria:

● No specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult people with suspected Long COVID can participate in this study. As the study is completely digital, there are no restriction in terms of living country.
  All the users of the Long COVID Companion app will be invited to participate in the study (by email or directly in the app). Recruitment will also be done by communications on social media, and by distributing study flyers in the waiting rooms of Long COVID consultations network. Participants to the PrediCOVID study who accepted to be recontacted will also be invited. Information regarding the study will also be disseminated to all people with Long COVID in the database of the Long COVID consultation network in Luxembourg.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue level | From enrollment until 24 months after
  Level of fatigue will be assessed regularly using a 0-5 likert scale. Participants will complete these questionnaires when they want during the follow-up.
Fatigue level | From enrollment until 24 months after
  Level of fatigue will be assessed regularly using FSS9 questionnaire. Participants will complete these questionnaires when they want during the follow-up.
Voice features | From inclusion until 24 months after
  * Source features (e.g., jitter, shimmer) reflecting the origin of voice production
  * Formant features (e.g., F1, F2, F3 frequencies, bandwidths) representing resonant frequencies of vocal and nasal tracts
  * Spectral features (e.g., centroid, MFCCs, flatness) capturing frequency distribution at specific moments
  * Prosody features (e.g., pitch, intensity, speech rate, pause duration) describing rhythm and intonation

CONTACTS AND LOCATIONS:
Locations (1):
- LIH, Strassen, Luxembourg

IPD SHARING:
Plan to Share IPD: No